CLINICAL TRIAL: NCT02115464
Title: A Phase II Study to Investigate a Combination of Metformin With Chemo-Radiotherapy in Patients With Locally Advanced Non-Small Cell Lung Cancer
Brief Title: Advanced Lung Cancer Treatment With Metformin and Chemo-Radiotherapy
Acronym: ALMERA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The accrual rate was not high enough to reach the target sample size.
Sponsor: Ontario Clinical Oncology Group (OCOG) (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OCOG-2014-ALMERA
Record Dates: First submitted 2014-04-14; First posted 2014-04-16 (Estimated); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Lung Cancer
Keywords: Metformin; Non-small cell lung cancer; Locally advanced; Chemo-radiotherapy; Lung cancer treatment
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metformin plus Chemo-radiotherapy (Experimental): Metformin orally 500 mg twice daily for the first week, 1500 mg a day in week 2 and 2000 mg a day at week 3 and then for a period of 12 months. Cisplatin-based chemotherapy with or without consolidation with standard radiotherapy of 60-63 Gy for 6 weeks.
  Interventions: Drug: Metformin plus Chemo-radiotherapy
- Chemo-radiotherapy (Active Comparator): Concurrent cisplatin based chemotherapy with or without consolidation and radiotherapy of 60-63 Gy for 6 weeks.
  Interventions: Radiation: Chemo-radiotherapy

INTERVENTIONS:
Drug: Metformin plus Chemo-radiotherapy — Metformin 2000 mg a day for 12 months plus cisplatin-based chemotherapy with or without consolidation with standard radiotherapy of 60-63 Gy for 6 weeks.
  Other Names: Metformin Hydrochloride
  Arms: Metformin plus Chemo-radiotherapy
Radiation: Chemo-radiotherapy — Cisplatin-based chemotherapy with or without consolidation with standard radiotherapy of 60-63 Gy for 6 weeks.
  Arms: Chemo-radiotherapy

SUMMARY:
ALMERA is a randomized, phase II, open label study in patients with locally advanced non-small cell lung cancer (NSCLC) which will compare standard radiotherapy plus concurrent chemotherapy with or without consolidation versus the same treatment plus concurrent Metformin continuing for 12 months. Metformin is a well tolerated and inexpensive drug that has the potential to improve cancer patient outcomes.

DETAILED DESCRIPTION:
This is a randomized, phase II, open label study in patients with locally advanced NSCLC which will compare standard RT (60-63 Gy for 6 weeks) plus concurrent Cisplatin-based chemotherapy (CRT) with or without consolidation (standard arm) vs the same CRT with or without consolidation plus treatment with Metformin concurrent with CRT and continuing for a total of 12 months (experimental arm). Ninety-four eligible and consenting patients will be randomized to one of the two treatment arms. Patients randomized to the experimental arm will receive Metformin (2000 mg/day) for a period of 12 months. Patients will be continuously evaluated for toxicity, will be assessed weekly at clinic visits during concurrent CRT treatment with or without consolidation and at follow up clinic visits at 3, 6, 9 and 12 months (from the date of randomization). Disease progression will be evaluated every 3 months for up to 12 months. All patients will be followed for up to 24 months (2 years) for survival.

The primary objective of this study is to determine the effect of Metformin on the proportion of patients free of disease progression at 12 months after initiation of drug treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age >/=18 to </= 80 years of age.
2. Unresected and pathologically (histologic) proven Stage 3a or Stage 3b NSCLC of adenocarcinoma, squamous cell, large cell or mixed histology, diagnosed within three months of study randomization.
3. Non-metastatic disease staged by: CT-chest and upper abdomen, brain MRI or contrast-enhanced CT within 12 weeks and physical examination and whole body FDG-PET/CT scan within 8 weeks prior to study randomization.

Exclusion Criteria:

1. Eastern Cooperative Oncology Group (ECOG) performance status >2.
2. More than 10% weight loss in the past 3 months.
3. Diabetic patient or anyone currently taking Metformin, insulin or other anti-hyperglycemic therapy.
4. Pulmonary Function Test (PFTs) (within the last 12 weeks) with Forced Expiratory Volume (FEV)1 < 1.2 litres per second or less than 50% of predicted.
5. Complete Blood Count (CBC) and biochemical renal and liver function profiles that do not permit chemotherapy treatment (as per institutional standard of care).
6. Fasting blood sugar levels of >/= 7.0 mmol per litre (within the last 12 weeks).
7. Prior systemic chemotherapy for lung cancer.
8. Prior radiotherapy that would overlap with the planned treatment area.
9. Prior invasive malignancy within the past 3 years (except non-melanomatous skin cancer non-invasive carcinoma in-situ of the breast, oral cavity or cervix).
10. Known Acquired Immune Deficiency Syndrome (AIDS).
11. Patients with increased risk for lactic acidosis:

    * severe congestive heart failure (NYHA: class III or IV),
    * history of metabolic acidosis,
    * alcoholic intake of > 3 drinks daily,
    * severe liver disease,
    * renal failure
12. Known hypersensitivity or allergy to Metformin.
13. Known pregnancy or lactating female patient.
14. Geographic inaccessibility for follow-up.
15. Inability to provide informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2014-12-17 (Actual); Primary Completion 2020-03-09 (Actual); Study Completion 2020-04-21 (Actual)

PRIMARY OUTCOMES:
Progression free survival | 12 months
  Progression free survival illustrates loco-regional disease control and freedom from distant metastasis

SECONDARY OUTCOMES:
Overall survival | 18-24 months
  Overall survival will be defined from the date of randomization until the date of death due to any cause.
Time to loco-regional progression | 18-24 months
  Time to loco-regional progression is defined from the date of randomization until the date of confirmed loco-regional progression
Distant progression-free survival | 18-24 months
  Distant progression-free survival is defined from the date of randomization until the date of distant progression, or death due to any cause.
Toxicities | 12 months plus 30 days
  The adverse event reporting period begins from the time of randomization and ends 30 days after the last treatment (concurrent chemo-radiotherapy plus or minus Metformin). Only adverse events assessed as Grade 3 or higher will be documented.

CONTACTS AND LOCATIONS:
Overall Officials: Theodoros Tsakiridis, MD, Principal Investigator — Juravinski Cancer Centre, Hamilton, Ontario, Canada
Locations (7):
- Canada (7):
  - Cross Cancer Institute, Edmonton, Alberta
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Juravinski Cancer Centre, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston General Hospital, Kingston, Ontario
  - Grand River Regional Cancer Centre, Kitchener, Ontario
  - Walker Family Cancer Centre - Niagara Health System, St. Catharines, Ontario
  - Montreal General Hospital - McGill, Montreal, Quebec

REFERENCES:
- [Derived] Tsakiridis T, Pond GR, Wright J, Ellis PM, Ahmed N, Abdulkarim B, Roa W, Robinson A, Swaminath A, Okawara G, Wierzbicki M, Valdes M, Levine M. Metformin in Combination With Chemoradiotherapy in Locally Advanced Non-Small Cell Lung Cancer: The OCOG-ALMERA Randomized Clinical Trial. JAMA Oncol. 2021 Sep 1;7(9):1333-1341. doi: 10.1001/jamaoncol.2021.2328. PMID 34323924